



## **Informed Consent Form**

## Assessing gastric emptying using spectroscopy

Study title: Non-invasive transcutaneous spectroscopy for the assessment of gut permeability (GutPerm)

IRAS Project ID: 242462

| Pa | tient Trial ID Number: | | | | |
|---|---|---|---|---|---|
| Na | nme of Principal Investigator: <u>D</u> i | r Alex Thompson | | | |
| Na | ame of patient to whom this ICF ap | oplies: | | | |
| | | | | Please | initial boxes: |
| 1. | I confirm that I have read and understand the Participant Information Sheet "Assessing gastric emptying using spectroscopy v4.1A 06-Mar-2019" for the above study and have had the opportunity to ask questions about the study and understand what is involved. | | | | |
| 2. | <ol> <li>I understand that my participation is voluntary and that I am free to withdraw at any time, without<br/>giving any reason, without my medical care or other legal rights being affected, and I understand<br/>that any remaining samples will be destroyed at my request, but data collected up to the point of<br/>my withdrawal may still be used.</li> </ol> | | | | |
| 3. | . I confirm that I have had sufficient time to consider if want to be included in the study. | | | | |
| 4. | I. I agree to allow information about me to be collected, analysed, reported and transferred to other approved collaborators within and outside the European Economic Area for healthcare and/or medical research purposes. I understand that my identity will remain anonymous. | | | | |
| 5. | I wish to be contacted by e-mail with a summary of the research findings once the study is complete. Your e-mail address will not be used for any other purpose. | | | | |
| | Contact e-mail: | | | | |
| | If you do <u>NOT</u> wish to be contacted regarding the study results, please put a line through all of point 5 above, do <u>NOT</u> leave a contact e-mail address and do <u>NOT</u> initial the box as indicated – you can still participate in the main trial. | | | | |
| 6. | I agree to take part in the study. | | | | |
| Ple | ease sign and date below. | | | | |
| Na | me of Subject | Signature | Date | | |
| <br>Na | me of Person taking consent | Signature | Date | <del></del> | |

1 copy for subject; 1 copy for Principal Investigator; 1 copy to be kept with hospital notes

IRAS ID: 242462